CLINICAL TRIAL: NCT04198922
Title: Acalabrutinib for Chronic Graft-Versus-Host Disease
Brief Title: Acalabrutinib for the Treatment of Chronic Graft Versus Host Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1006135; NCI-2019-06980 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 8801 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-12-05; First posted 2019-12-13 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Moderate-Severe Chronic Graft Versus Host Disease; Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — acalabrutinib; benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (acalabrutinib) (Experimental): Patients receive acalabrutinib 100 mg PO BID on days 1-28. Treatment repeats every 28 days for up to 6 cycles with an option to continue for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Acalabrutinib; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: 1420477-60-6; ACP-196; Benzamide; Bruton Tyrosine Kinase Inhibitor ACP-196
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well acalabrutinib works in treating patients with chronic graft versus host disease. Acalabrutinib may be an effective treatment for graft-versus-host disease caused by a stem cell transplant.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive acalabrutinib orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 6 cycles with an option to continue for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age
* Moderate-severe chronic GVHD, diagnosed per the 2014 National Institutes of Health (NIH) criteria
* Progression or recurrence of active chronic GVHD signs/symptoms after treatment with steroids
* Karnofsky performance status >= 70%
* Woman of childbearing potential (WOCBP) who are sexually active must use highly effective methods of contraception during treatment and for 2 days after the last dose of acalabrutinib
* Men must refrain from sperm donation during the study
* Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information

Exclusion Criteria:

* Hospitalization for evaluation or management of an infection within the last 8 weeks
* Change in immunosuppressive regimen within the 2 weeks prior to enrollment
* Noncompliance
* Treatment of chronic GVHD with ibrutinib
* Received any investigational drug within 30 days or 5 half-lives (whichever is shorter) before first dose of study drug
* Recurrent or prior malignancy (or any other malignancy that requires active treatment), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for >= 2 years
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 or 4 cardiac disease as defined by the New York Heart Association functional classification. Subjects with controlled, asymptomatic atrial fibrillation during screening can enroll on study
* Has difficulty with or is unable to swallow oral medication, or has significant gastrointestinal disease that would limit absorption of oral medication
* Received a live virus vaccination within 28 days of first dose of study drug
* Known history of infection with human immunodeficiency virus (HIV)
* Uncontrolled, active significant infection (e.g., bacterial, viral, fungal or progressive multifocal leukoencephalopathy)
* Known history of drug-specific hypersensitivity or anaphylaxis to study drug (including active product or excipient components)
* Active bleeding, history of bleeding diathesis (e.g., hemophilia or von Willebrand disease)
* Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura)
* Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer
* Requires warfarin or equivalent vitamin K antagonist
* History of significant cerebrovascular disease or event, including stroke or intracranial hemorrhage, within 6 months before the first dose of study drug
* Major surgical procedure within 30 days of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug
* Subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HBsAg) positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded
* Child-Pugh score of C for hepatic impairment
* Total bilirubin > 2 mg/dL or alanine aminotransferase (ALT) > 2 x upper limit of normal, unless abnormalities are due to liver GVHD, in which case total bilirubin > 3 mg/dL or ALT 5 x upper limit of normal are exclusions
* Absolute neutrophil count < 1.0 x 10^9/L or use of myeloid growth factors within the past 2 weeks
* Platelet count < 50 x 10^9/L or platelet transfusion or thrombomimetic agent within the past 2 weeks
* Glomerular filtration rate < 50 mL/min/1.73 m^2
* Breastfeeding or pregnant
* Concurrent participation in another clinical trial and receiving a non-Food and Drug Administration (FDA) approved medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Best response (complete and partial response [CR + PR]) | Within the first 6 months of treatment when the best response rate is known for each patient
  The composite outcome of CR and PR, calculated according to the proposed response definitions of the 2014 National Institutes of Health Consensus Conference. Exact 95% confidence intervals (CI) will be calculated for the objective response rate using the Clopper and Pearson method. Will also compare the observed best ORR with the published efficacy of ibrutinib (67%) and provide the 95% CI for the difference.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days following the last dose of acalabrutinib
  Defined as grade 3 and above according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 and all serious AEs (SAEs) described for the population receiving at least one dose of acalabrutinib at least from the time of consent through the safety follow-up period. Any AE/SAE at least possibly related to acalabrutinib therapy will be reported for the duration of the study.
Duration of response (DOR) | From the date the PR is documented until loss of the response or start of another systemic immunosuppressive treatment for chronic graft versus host disease (GVHD), whichever occurs first, assessed up to 3 years
  Will be described for the group achieving at least a PR, defined as the number of weeks the subject maintains a PR or CR. Will be estimated using the Kaplan-Meier method. Approximate 95% CIs for median DOR will be computed using the formula proposed by Brookmeyer and Crowley.
Change in patient-reported outcomes: Lee Chronic GVHD Symptom Scale score | Baseline up to 3 years
  Will be assessed by the Lee Chronic GVHD Symptom Scale score. Scores will be calculated based on published algorithms with absolute changes and clinically meaningful changes described for the population as a whole and based on CR + PR versus stable disease (SD) + mixed response (MR) + progressive disease (PD).
Change in patient-reported outcomes: Patient-Reported Outcomes Measurement Information System-29 | Baseline up to 3 years
  Will be assessed by the Patient-Reported Outcomes Measurement Information System-29. Scores will be calculated based on published algorithms with absolute changes and clinically meaningful changes described for the population as a whole and based on CR + PR versus stable disease (SD) + mixed response (MR) + progressive disease (PD).
Failure-free survival | At 6 months and 1 year
  Will be defined as the duration of relapse-free survival without adding any other systemic treatment for chronic GVHD. Will be estimated with the composite event of death from any cause, relapse and addition of secondary immune suppressive agents using the Kaplan-Meier method. Systemic immune-suppressive agents include orally or intravenously administered systemically active immune-suppressive drugs, as well as procedures including extra-corporeal photopheresis.
Organ-specific response rates | Up to 3 years
  Response rates by organ will also be calculated and reported as ORR (CR+PR) versus all other categories (SD, PD, MR).

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lee, MD, MPH, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (6):
- United States (6):
  - Moffitt Cancer Center, Tampa, Florida
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT04198922/ICF_000.pdf